CLINICAL TRIAL: NCT02895126
Title: Assessment of the "Appui Parental": A Program of Early Support to Parenthood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9237
Record Dates: First submitted 2016-08-30; First posted 2016-09-09 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Infant Development
Keywords: vulnerable family

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Appui Parental" program (44 cases) (Experimental)
  Interventions: Behavioral: "Appui Parental" program
- Regular parental support (44 cases) (Other): Usual intervention
  Interventions: Behavioral: Regular parental support

INTERVENTIONS:
Behavioral: "Appui Parental" program
  Arms: "Appui Parental" program (44 cases)
Behavioral: Regular parental support
  Arms: Regular parental support (44 cases)

SUMMARY:
In so-called at risk families, the child-parent attachment relationship is more difficult to set up and this can be a barrier to social and emotional development of young children. To help parents build and sustain this relationship, and to prevent child development disorders, many parenting programs have been created, usually with frequent home visits by early childhood professionals. In France, therapeutic interventions at home are little used and they are not evaluated.

In Montpellier, an action of this type has been conducted since 2001 by the "Conseil Départemental de l'Hérault" in collaboration with the University Hospital of Montpellier including, in addition to home visits, supervision of professionals: the Appui Parental Program.

Before extending this action to other areas of Herault, the "Conseil Départemental de l'Hérault", the "Abri Languedocien" and the University Hospital of Montpellier are conducting an assessment to know the effectiveness of the program for families under care.

This 3-year multicenter prospective study includes 88 children aged 1 to 20 months from families meeting vulnerability criteria previously defined, 44 benefiting Appui Parental program (experimental group) and 44 benefiting a regular support (control group).

A paediatric examination on the basis of the Denver scale, parental questionnaires, questionnaires to professionals and an a video of infant-parent interactions are used. The data, collected at baseline and 18 months later, will be compared.

DETAILED DESCRIPTION:
Objective: the main objective of this study is to determine the efficiency of Appui Parental program by evaluating its impact on the development of children aged from 0 to 3 years. The secondary objectives are to study the effects of the intervention on: the mother-child interactions, the degree of therapeutic alliance between parent and professionals, the parenting skills feeling, perceived social support, anxiety and depression of parents, frequency of legal interventions (placements, educational measures). An assessment of stress among professionals involved in the study and evaluation of the therapeutic alliance with families will also be conducted to assess the effectiveness of the supervision included in the program.

Hypothesis: Scores on Symptom Check List after 18 months of follow up will be significantly higher in subjects who benefited the Appui Parental program compared to subjects with conventional parental support. Similarly, it is expected that other developmental assessments of children have the best results in the Appui Parental Program group than in the control group. Finally, it is assumed that the mother-child interactions, the parenting skills feeling, and the therapeutic alliance between parent and professional are better in the Appui Parental program than in the control group.

ELIGIBILITY:
Inclusion Criteria:

* family with child between 1 and 20 months of age and with parents eligible to parental support,
* written informed consent signed by both parents or 1 legal guardian,
* vulnerability criteria with difficulties to meet the needs of their child,
* family affiliated to social security.

Exclusion Criteria:

* mother having delusional psychosis,
* family whose child is in danger and needs an immediate protective measure,
* ongoing justice procedure for the child,
* family with impossibility to follow-up during 18 months,
* non French-speaking parents.

Ages: 1 Month to 20 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Symptom Check-List (SCL) score variation | up to 18 months

SECONDARY OUTCOMES:
Child Behavior Check-List (CBCL) score variation | up to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France